CLINICAL TRIAL: NCT00663715
Title: Anatomical Description of the Sciatic Nerve Via a Lateral Mid-Thigh Approach Using Ultrasound
Brief Title: Ultrasound Description of the Sciatic Nerve
Status: Withdrawn | Type: Observational
Why Stopped: No subjects were enrolled. Sciatic blocks infrequently used for pain control.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-02-5808
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2010-04

CONDITIONS: Sciatic Nerve AH; Peripheral Nerves US
Keywords: Sciatic Nerve; Peripheral Nerve Block; Lower extremity surgery; Local Anesthesia; Ultrasound guided nerve blocks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Pediatric Patients of ages 11-17
  Interventions: Other: Observation of the Sciatic Nerve

INTERVENTIONS:
Other: Observation of the Sciatic Nerve — Ultrasound will be used to determine the location of the Sciatic Nerve using a lateral mid-thigh approach.
  Other Names: Sciatic Nerve location; Peripheral Nerve Blocks

SUMMARY:
Sciatic nerve blocks are frequently used for anesthesia or analgesia for surgery of the lower legs. Currently, if ultrasound is used to find the sciatic nerve, the leg must be raised to locate the nerve with the ultrasound probe on the back of the thigh. In pediatric surgery, the patients are anesthetized (asleep) before the block is given. It is difficult for one person to administer the sciatic nerve block using this method. We would like to identify the sciatic nerve using ultrasound on the side of the thigh and its location to the adjacent structures.

DETAILED DESCRIPTION:
The sciatic nerve block is frequently used for anesthesia or analgesia for surgery of the lower extremities. Ultrasound-guided sciatic nerve blocks performed at the lateral mid-femoral level have been successfully described with subjects in the supine position and the lower limb elevated in order to accommodate the ultrasound probe against the posterior aspect of the thigh. In the pediatric setting in which nerve blocks are commonly performed with the patient anesthetized rather than awake, we find this technique to be unwieldy as a single-operator technique. Using a more ergonomic approach that has not been previously described, we plan to identify and describe the sciatic nerve with the ultrasound positioned against the lateral aspect of the thigh. We hope to describe the appearance of the sciatic nerve and its location in relation to adjacent anatomic structures using this modified approach.

This a prospective cross-sectional study of 40 pediatric subjects 11-17 years of age. Three ultrasound images of the sciatic nerve will be obtained via the lateral mid-thigh approach in 40 pediatric patients scheduled to undergo sciatic nerve block - the first image prior to placement of the block, the second after the nerve is located by the stimulating needle and the third after the injection of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 11 to 17 years old.
2. Patients undergoing lower extremity surgery who are scheduled to have a sciatic nerve block as part of the anesthetic.
3. Parental/guardian permission (verbal consent) and child assent. Note: if you record ANY PHI, you will need to obtain written consent since HIPAA requires written authorization for use of PHI.

Exclusion Criteria:

None

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to describe the appearance of the sciatic nerve and its location in relation to adjacent anatomic structures using ultrasound from the lateral mid-thigh position. | 10 minutes

SECONDARY OUTCOMES:
A secondary objective is to describe correlations between any of the measured variables and the patient's mid-thigh circumference or weight. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Arjunan Ganesh, MBBS, Principal Investigator — Children's Hospital of Philadelphia

REFERENCES:
- [Background] Karmakar MK, Kwok WH, Ho AM, Tsang K, Chui PT, Gin T. Ultrasound-guided sciatic nerve block: description of a new approach at the subgluteal space. Br J Anaesth. 2007 Mar;98(3):390-5. doi: 10.1093/bja/ael364. PMID 17307781